CLINICAL TRIAL: NCT00721162
Title: A Phase 2, Non-randomized, Open-label, Multicenter Study of IMC-1121B in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: Study of Ramucirumab in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13923; 2007-006717-17 (EudraCT Number); CP12-0711 (Other: ImClone Systems); I4T-IE-JVBR (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-07-21; First posted 2008-07-23 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian Cancer,; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ramucirumab (Experimental)
  Interventions: Biological: Ramucirumab

INTERVENTIONS:
Biological: Ramucirumab — Participants will receive ramucirumab at 8 milligrams/kilogram (mg/kg) administered over 1 hour every other week (every 14 days). Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met.
  Other Names: IMC-1121B

SUMMARY:
The purpose of this study is to determine if ramucirumab given as monotherapy is effective in the treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma.

DETAILED DESCRIPTION:
Current chemotherapies used to treat ovarian cancer participants include doxorubicin, topotecan, and paclitaxel, to mention a few. Doxorubicin was studied in ovarian cancer participants that were refractory to paclitaxel and platinum-based chemotherapy agents. Inhibition of angiogenesis is considered a promising approach to the treatment of cancer. Vascular endothelial growth factor (VEGF) is an important regulator of angiogenesis and is likely an important therapeutic target in persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. VEGF is overexpressed in ovarian tissue and may be the most important single tumor angiogenic factor. Phase 1 studies currently nearing completion with ramucirumab have demonstrated safety and tolerability at clinically relevant doses, with preliminary evidence of clinical efficacy in ovarian cancer participants. Therefore, ImClone Systems plans to conduct a Phase 2 trial to assess the safety and efficacy of ramucirumab in participants with platinum-refractory persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet the following criteria to be enrolled in this study:

1. The participant has recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. Histologic documentation of the original primary tumor is required via a pathology report
2. The participant has at least one unidimensional-measurable target lesion [≥ 2 centimeter (cm) with conventional techniques, or ≥ 1 cm by spiral computed tomography (CT) or magnetic resonance imaging (MRI)], as defined by Response Evaluation Criteria in Solid Tumors (RECIST). Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
3. The participant has recovered to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 3.0 (NCI-CTCAE v3.0) from the effects of recent surgery, radiotherapy, chemotherapy, hormonal therapy, or other targeted therapies for ovarian cancer, with the exception of alopecia or peripheral neuropathy (which must have resolved to Grade ≤ 2). Any other prior therapy directed at the malignant tumor must be discontinued at least three weeks prior to the first dose of study medication, or hormonal therapy discontinued at least one week prior to the first dose of study medication. Continuation of hormone replacement therapy is permitted
4. The participant has completed at least one platinum-based chemotherapeutic regimen for management of primary disease, and must have at least one of the following: a platinum-free interval of < 12 months after the final dose of primary platinum-based therapy, progression during platinum-based therapy, or persistent disease after platinum-based therapy
5. The participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1 at study entry
6. The participant has adequate hematological functions [absolute neutrophil count (ANC) ≥ 1200 cells/microliter (uL), hemoglobin ≥ 9 grams/deciliter (g/dL), and platelets ≥ 100,000 cells/uL]
7. The participant has adequate hepatic function [bilirubin ≤ 1.5 times the upper limit of normal (ULN); aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 3.0 times ULN, or ≤ 5.0 times ULN if the transaminase elevation is due to liver metastases]
8. The participant has adequate renal function [serum creatinine ≤ 1.5 x ULN or creatinine clearance (measured or calculated) ≥ 60 milliliters/minute (mL/min)]
9. The participant's urinary protein is ≤ 1+ on dipstick or routine urinalysis (UA). If urine dipstick or routine analysis indicated ≥ 2+ proteinuria, then a 24-hour urine must be collected and must demonstrate < 1000 milligrams (mg) of protein in 24 hours to allow participation in the study
10. The participant has adequate coagulation function, as defined by international normalized ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 1.5 X ULN if not receiving anticoagulation therapy. Participants on full-dose anticoagulation must be on a stable dose of oral anticoagulant or low molecular weight heparin, and if on warfarin must have therapeutic INR and have no active bleeding (defined as within 14 days of first dose of study medication) or pathological condition that carries a high risk of bleeding (example, tumor involving major vessels or known varices)
11. For participants who have received anthracycline therapy, the left ventricular ejection fraction (LVEF) must be within normal institutional range by a pretreatment echocardiogram or multigated acquisition (MUGA) scan
12. If sexually active, the participant is post-menopausal, surgically sterile, or using effective contraception in the opinion of the investigator
13. The participant is ≥ 18 years of age
14. The participant has a life expectancy of ≥ 3 months
15. The participant is able to provide informed written consent and is amenable to compliance with protocol schedules and testing

Exclusion Criteria:

1. The participant has a concurrent active malignancy, other than adequately treated nonmelanomatous skin cancer or other noninvasive carcinoma or in situ neoplasm. A participant with previous history of malignancy is eligible provided that she has been disease-free for > 3 years
2. The participant has received a noncytotoxic regimen (usually called targeted therapy such as bevacizumab) for recurrent or persistent disease. (Participants may have received a noncytotoxic regimen as primary treatment.)
3. The participant has received radiotherapy for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within 3 weeks (21 days) prior to the first dose of study medication
4. The participant has received prior radiotherapy to any portion of the abdominal cavity or pelvis other than for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last 3 years. [Prior radiation for localized cancer (for example, of the breast, head and neck, or skin) is permitted, provided that it was completed > 3 years prior to the first dose of study medication, and the participant remains free of recurrent or metastatic disease.]
5. The participant has received prior chemotherapy for any abdominal or pelvic tumor, other than for the treatment of ovarian, fallopian tube, or primary peritoneal cancer < 3 years prior to the first dose of study medication. Prior adjuvant chemotherapy for localized breast cancer is permitted, provided that it was completed >3 years prior to the first dose of study medication, and that the participant remains free of recurrent or metastatic disease
6. The participant has undergone major abdominal surgery within 4 weeks (28 days) prior to first dose of study medication
7. The participant has a suspected impending bowel obstruction, based on clinical or radiographic criteria
8. The participant has received any hormonal therapy directed at the malignant tumor discontinued therapy within 1 week (7 days) prior to first dose of study medication
9. The participant has received any other prior therapy directed at the malignant tumor, including immunologic agents, within 3 weeks (21 days) prior to first dose of study medication
10. The participant has received previous treatment with ramucirumab
11. The participant has participated in clinical trials of experimental agents within 4 weeks (28 days) prior to first dose of study medication
12. The participant has a history of uncontrolled hereditary or acquired bleeding or thrombotic disorders
13. The participant has an ongoing or active infection requiring systemic antibiotics, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, myocardial infarction < 6 months, Grade ≥ 2 peripheral vascular disease, poorly controlled hypertension despite standard medical management poorly controlled thrombotic or hemorrhagic disorder, psychiatric illness or social situations that would limit compliance with study requirements, or any other serious uncontrolled medical disorders in the opinion of the investigator
14. The participant has any history of brain metastases or leptomeningeal disease. Screening for central nervous system (CNS) involvement for testing asymptomatic participants is not required
15. The participant has known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
16. The participant is pregnant [confirmed by serum beta human chorionic gonadotropin (β-HCG) test] or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (11):
  - ImClone Investigational Site, Hollywood, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Chicago, Illinois
  - ImClone Investigational Site, Marrero, Louisiana
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Baltimore, Maryland
  - ImClone Investigational Site, Boston, Massachusetts
  - ImClone Investigational Site, Rochester, Minnesota
  - ImClone Investigational Site, Oklahoma City, Oklahoma
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Seattle, Washington
- United Kingdom (2):
  - ImClone Investigational Site, London
  - ImClone Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Penson RT, Moore KM, Fleming GF, Braly P, Schimp V, Nguyen H, Matulonis UA, Banerjee S, Haluska P, Gore M, Bodurka DC, Hozak RR, Joshi A, Xu Y, Schwartz JD, McGuire WP. A phase II study of ramucirumab (IMC-1121B) in the treatment of persistent or recurrent epithelial ovarian, fallopian tube or primary peritoneal carcinoma. Gynecol Oncol. 2014 Sep;134(3):478-85. doi: 10.1016/j.ygyno.2014.06.029. Epub 2014 Jul 10. PMID 25016924

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 73 participants signed informed consent.
Groups:
- Ramucirumab: Ramucirumab at 8 milligrams/kilogram (mg/kg) administered intravenously over 1 hour every other week (every 14 days) of a 28-day cycle.
Period: Overall Study
Arm/Group | Ramucirumab
Started | 60
Received Any Amount of Study Drug | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received any amount of study drug.
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5
  White | 52
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 56
  United Kingdom | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival at 6 Months (PFS-6)
Description: Data presented are the percentage of participants without progressive disease (PD) or death from any cause at 6 month after first dose. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PD is ≥20% increase in sum of longest diameter of target lesions and/or unequivocal progression of non-target lesion and/or new lesion.
Time Frame: First Dose to 6 Months
Population: All participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
percentage of participants | 25.0 [14.7 to 37.9]

2. Primary Outcome: Objective Response Rate (ORR): Percentage of Participants With Complete Response (CR) and Partial Response (PR)
Description: Objective response is confirmed complete response (CR) + partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesion. ORR is calculated as a total number of participants with CR or PR from the start of study treatment until disease progression/recurrence or the start of new therapeutic anticancer treatment, whichever occurred first, divided by the total number of participants treated, then multiplied by 100.
Time Frame: First dose to date of objective progressive disease /death or new anti-cancer therapy up to 34.6 months
Population: All participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
percentage of participants | 5.0 [1.0 to 13.9]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: Defined as the time from date of first dose to the first observation of progression of disease (PD) or death due to any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PD is ≥20% increase in sum of longest diameter of target lesions and/or unequivocal progression of non-target lesion and/or new lesion. For participants who had no PD or death or had started new therapeutic anticancer treatment, PFS was censored at their last radiographic tumor assessment.
Time Frame: First dose to measured progressive disease or death due to any cause up to 34.6 months
Population: All participants who received any amount of study drug. The number of participants censored was 11.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
months | 3.5 [2.3 to 5.3]

4. Secondary Outcome: Overall Survival at 1 Year (OS-1)
Description: Data presented are the percentage of participants surviving at least 12 months after first dose based on Kaplan Meier Method.
Time Frame: First dose to 12 months
Population: All participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
percentage of participants | 48.0 [34.9 to 59.9]

5. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from first dose to the date of death due to any cause. For participants who were alive or were lost to follow-up, overall survival was censored on the last date the participant was known to be alive.
Time Frame: First dose to death due to any cause up to 43.9 months
Population: All participants who received any amount of study drug. The number of participants censored was 12.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
months | 11.1 [8.3 to 17.0]

6. Secondary Outcome: Summary Listing of Participants Reporting Drug-Related Treatment-Emergent Adverse Events
Description: Data presented are the number of participants who experienced treatment-emergent adverse events (TEAE), serious adverse events (SAE), Grade 3 or 4 TEAE, or adverse events (AE) leading to discontinuation of treatment that were considered to be related to ramucirumab. A summary of SAEs and other nonserious AEs, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: First dose to 30 months
Population: All participants who received any amount of study drug.
Measure: Number; unit: participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 60
participants
  Related TEAE | 56
  Related SAE | 10
  Related Grade 3 or 4 TEAE | 21
  Related AE leading to discontinuation | 4

ADVERSE EVENTS:
Description: Deaths due to progressive disease are not considered adverse events (AE). Four deaths due to progressive disease were recorded by the investigator as serious AEs (SAE) and are captured in the SAE summary.
Arm/Group | Ramucirumab
Serious Adverse Events (participants affected / at risk) | 22/60
Other Adverse Events (participants affected / at risk) | 58/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (5)
Vomiting (Gastrointestinal disorders) | 1 (1)
Abscess sterile (General disorders) | 1 (1)
Hernia obstructive (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Peritonitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Expired drug administered (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5)
Neuralgia (Nervous system disorders) | 1 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=60)
Anaemia (Blood and lymphatic system disorders) | 11 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (20)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 12 (14)
Abdominal pain lower (Gastrointestinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 13 (15)
Diarrhoea (Gastrointestinal disorders) | 21 (41)
Dyspepsia (Gastrointestinal disorders) | 6 (8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 6 (10)
Nausea (Gastrointestinal disorders) | 26 (38)
Stomatitis (Gastrointestinal disorders) | 11 (15)
Vomiting (Gastrointestinal disorders) | 20 (31)
Chills (General disorders) | 5 (8)
Fatigue (General disorders) | 41 (72)
Oedema peripheral (General disorders) | 16 (23)
Pyrexia (General disorders) | 8 (11)
Nasopharyngitis (Infections and infestations) | 4 (6)
Sinusitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (5)
Urinary tract infection (Infections and infestations) | 13 (19)
Alanine aminotransferase increased (Investigations) | 4 (7)
Aspartate aminotransferase increased (Investigations) | 4 (11)
Weight decreased (Investigations) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 12 (16)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (13)
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11)
Dizziness (Nervous system disorders) | 7 (8)
Dysgeusia (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 43 (72)
Insomnia (Psychiatric disorders) | 7 (7)
Proteinuria (Renal and urinary disorders) | 8 (10)
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Flushing (Vascular disorders) | 5 (6)
Hypertension (Vascular disorders) | 16 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.